CLINICAL TRIAL: NCT03888638
Title: Search for the Clinical Significance of Tumor-associated Macrophages in Patients With Colorectal Liver Metastases
Brief Title: The Role of Tumor-associated Macrophages in Colorectal Liver Metastases
Status: Completed | Type: Observational
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Matteo Donadon, Assistant Professor of Surgery, Humanitas Clinical and Research Center
Other Study IDs: TAMs in CLM
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Liver Metastases; Colorectal Cancer; Liver Metastases; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Specimens from liver resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hepatectomy — Removal of a part of the liver because of tumor
  Other Names: Liver resection

SUMMARY:
Colorectal cancer is a major cause of mortality worldwide. Most patients develop colorectal liver metastases (CLM), and for such patients hepatectomy combined with chemotherapy may be curative. Nevertheless, in the era of precision medicine there is a critical need of prognostic markers to cope with the heterogeneity of CLM patients. Tumor-associated macrophages (TAMs) pave the way to tissue invasion and intravasation providing a nurturing microenvironment formetastases. The quantification of immune landscape of tumors has provided novel prognostic indicators of cancer progression, and the quantification of TAMs might explain the heterogeneity of CLM patients. Here, we will investigate the development of a new diagnostic tool based on TAMs with the aim to define the causative role of TAMs in CLM patients. This will open new clinical scenarios both for the diagnosis, therapy and prognosis, leading to the refinement of the therapeutic output in a personalized medicine perspective.

DETAILED DESCRIPTION:
Some preliminary data produced by the research team from Humanitas Clinical and Research Center in Milan (ITALY) have shown that TAMs in CLM are heterogeneous and that their diversity can be distinguished based on their morphology and functionality. Therefore, TAMs may represent an additional tool in the definition of the biology and prognosis of CLM patients. This preliminary finding provides us with the rationale to undertake a prospective study on a large series of CLM patients surgically resected by our unit aimed at validating the promisingcorrelation between different TAMs phenotypes and patients prognosis. The characterization of the diversity of TAMs in CLM will be refined using state of the art technology, including multi-parametric flow cytometry, single cell RNA sequencing (scRNA-seq) transcriptional profiling, metabolomic, and proteomic analyses. The expected findings will allow us to develop a new diagnostic tool based on TAMs features, which will open the way to new criteria for patient stratification and for the design of new targeted therapies in a personalized medicine perspective.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal liver metastases undergoing hepatectomy
* Full clinical, surgical, pathological and follow-up data
* Availability of tissues for the analysis

Exclusion Criteria:

* Missing (any) data
* Combination of radiofrequency or microwave ablation plus surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by colorectal liver metastases treated by hepatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Survival | From date of surgery until the date of first documented progression or date of death from any cause, which ever came first assessed up to 72 months]
  Analysis of survival after hepatic resection for colorectal liver metastases according with the tumor-associated macrophages characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Donadon, MD, PhD, Principal Investigator — Humanitas University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costa G, Sposito C, Soldani C, Polidoro MA, Franceschini B, Marchesi F, Nasir FD, Virdis M, Vingiani A, Leo A, Di Tommaso L, Kotha S, Mantovani A, Mazzaferro V, Donadon M, Torzilli G. Macrophage morphology and distribution are strong predictors of prognosis in resected colorectal liver metastases: results from an external retrospective observational study. Int J Surg. 2023 May 1;109(5):1311-1317. doi: 10.1097/JS9.0000000000000374. PMID 37037585